CLINICAL TRIAL: NCT00961506
Title: Prospective Evaluation of Laparoendoscopic Single Site Versus Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-08-145a
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Gallbladder Disease
Keywords: cholecystectomy; gallbladder; laparoscopy; laparoendoscopic
MeSH Terms: conditions — Gallbladder Diseases | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LESS cholecystectomy (Experimental): LESS cholecystectomy
  Interventions: Procedure: LESS cholecystectomy
- Laparoscopic cholecystectomy (Active Comparator): Laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: LESS cholecystectomy — LESS cholecystectomy
  Arms: LESS cholecystectomy
Procedure: Laparoscopic cholecystectomy — laparoscopic cholecystectomy
  Arms: Laparoscopic cholecystectomy

SUMMARY:
Laparoendoscopic single site cholecystectomy is associated with better cosmetic results and recovery compare to laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* gallbladder disease Age: 18-99

Exclusion Criteria:

* intolerance to laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Body image scale | 1 months

SECONDARY OUTCOMES:
pain VAS | 10 days
Analgesic requirement
time to return to work
scar scale | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Bucher, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland